CLINICAL TRIAL: NCT02857101
Title: The Ratio of Ascites Calprotectin to Total Protein is a Diagnostic and Prognostic Marker for Spontaneous Bacterial Peritonitis in Liver Cirrhosis
Brief Title: Calprotectin for Rapid Diagnostic Infection Spontaneous of Ascites
Acronym: Ca-DRISLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: BÜHLMANN Laboratories (Unknown)
Responsible Party: Sponsor
Other Study IDs: P/2015/243
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Rapid Diagnosis of Spontaneous Infection of Ascitic Fluid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: dosage of calprotectin

SUMMARY:
The prognosis of spontaneous bacterial peritonitis (ISLA) remains a serious complication of cirrhosis. Rapid diagnosis of ISLA is a key issue for improving the prognosis. The determination of calprotectin in ascites, used for the diagnosis of infection of ascitic liquid, could allow the diagnosis in a very short time (about 30 minutes). To date, the determination of calprotectin in ascites was not evaluated properly. The investigators would thus evaluate the interest of the determination of calprotectin in ascites for the rapid diagnosis of ISLA in cirrhotic patients, like you, hospitalized for decompensation of their disease. The main purpose of this pilot study will determine the optimal threshold calprotectin in ascites for diagnosis of ISLA.

DETAILED DESCRIPTION:
The occurrence of ascites in cirrhotic patients is a frequent event (about half of these patients developed ascites after 10 years of evolution) and marks an evolutionary turning point in the natural history of cirrhosis (30% survival at 5).

The spontaneous bacterial peritonitis (ISLA) is the leading infectious complication cirrhotic patient (prevalence of 10-30%). Half of these ISLA are already present on admission of the patient and over 20% of these infections are totally asymptomatic. The delay processing of ISLA causes heavy mortality. Even when antibiotic treatment is started immediately after the diagnosis of ISLA, in-hospital mortality remains high (about 20%) and mainly related to the development of severe sepsis, septic shock and hepatorenal syndrome; the medium-term prognosis remains severe as also survival after an episode of ISLA is 30-50% at 1 year. Therefore, the surviving patients with a first episode of ISLA are candidates for liver transplantation. Given the major prognostic implications and the asymptomatic nature of these infections, examination of ascites with neutrophil count (ANC) and bacteriological cultures still recommended during any puncture, which increases support. This is why clinicians are sensitive to processes that simplify the diagnosis of ISLA or make it faster.

The measurement of calprotectin in ascites could be of major interest for the rapid diagnosis of ISLA. It is a glycoprotein of 36 KDa fixing calcium and zinc, synthesized by neutrophils (where it represents 60% of the soluble proteins from the cytosol) as well as monocytes and macrophages in the lower concentration. It has anti-bacterial and anti-fungal, immunomodulatory and pro-apoptotic. Its synthesis is increased in case of inflammation and its rate reflects, in inflammatory bowel disease, the severity of the inflammation of the bowel wall. Fecal calprotectin allows to discriminate inflammatory bowel disease (IBD) functional impairment of the gastrointestinal tract (irritable bowel syndrome) in symptomatic patients and also seems more powerful than other non-specific markers of inflammation (CRP, sedimentation rate, leukocytosis) to make this distinction; again, this biological marker allows therapeutic monitoring for patients with IBD.

The reference technique proposed by the laboratory for assaying BÜHLMANN calprotectin is a quantitative ELISA in a stool sample or ascites but the Quantum Blue® Reader offers a faster quantitative measure (in 12 minutes). It consists of a sandwich immunoassay including the speed could be advantageously used for the diagnosis of ISLA. However, few studies have evaluated the assay of plasma calprotectin or in ascites in cirrhotic patients. A high plasma concentration of calprotectin could have a prognostic value in alcoholic cirrhosis, as a high concentration of calprotectin in ascites in decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years
* Presence of ascites due to cirrhosis
* Hospitalization for a complication of cirrhosis (first or recurrent ascites ascites decompensation requiring prolonged hospitalization, gastrointestinal bleeding, encephalopathy, etc ...).

Exclusion Criteria:

* Patients with ascites admitted to the hospital for a suspected infection and receiving an antibiotic for more than 12 hours (patients with antibiotic prophylaxis with norfloxacin with a clinical suspicion of ISLA will be included in the study (there may be in this case ISLA germs resistant to quinolones).
* Outpatient hospital to perform paracentesis evacuative
* Chylous ascites,
* Hemorrhagic Ascites
* Ascites not related to portal hypertension (peritoneal carcinomatosis, pancreatic ascites, tuberculosis, etc ...)
* comatose patients under guardianship or does not have all their mental faculties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cirrhotic patients over 18 years, with ascites and hospitalized for complications of their cirrhosis: ascites decompensation first or recurrent ascites requiring prolonged hospitalization (> 2 days), gastrointestinal bleeding, encephalopathy, etc.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Measurement of the calprotectin level in ascitic fluid with Quantum Blue® Reader | 18 months
  Establish an optimal threshold calprotectin in ascites for diagnosis of ISLA and evaluate the performance of calprotectin in ascites in cirrhotic patients with ascites due to portal hypertension only.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Besançon, Besançon, France